CLINICAL TRIAL: NCT04963361
Title: A Survey of Fear of Exercise and Its Influencing Factors in Patients After Total Knee Arthroplasty
Brief Title: Study on Fear of Movement After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021182
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fear of movement group: The score of fear of movement scale was more than 37
  Interventions: Other: patients were exposed to fear of movement
- non-fear of movement group: The score of fear of movement scale was no more than 37
  Interventions: Other: patients were not exposed to fear of movement

INTERVENTIONS:
Other: patients were exposed to fear of movement — Patients completed the questionnaires independently
  Groups: fear of movement group
Other: patients were not exposed to fear of movement — Patients completed the questionnaires independently
  Groups: non-fear of movement group

SUMMARY:
Total knee arthroplasty is one of the effective methods for the treatment of end-stage osteoarthritis. Postoperative rehabilitation exercise is an important method for the recovery of knee joint function. Exercise fear refers to an enlarged psychological phenomenon that patients are afraid of sports leading to injury, which is not conducive to the functional exercise of patients and hinders the recovery of knee joint function

DETAILED DESCRIPTION:
Object: the purpose of this study is to investigate the occurrence of fear of movement after total knee arthroplasty and analyze its influencing factors, so as to provide theoretical basis for reducing the occurrence of fear of movement after total knee arthroplasty, promoting the rehabilitation exercise of patients and promoting the recovery of knee joint function.

In this study, 121 patients with total knee arthroplasty were investigated by questionnaire, including general demographic data, sports fear scale, anxiety and depression scale, self-efficacy scale and so on. Multivariate logistic regression was used to analyze the influencing factors of postoperative fear of exercise.

ELIGIBILITY:
Inclusion Criteria:

（1） meeting the criteria of knee arthritis established by American Society of rheumatology （ 2) Total knee arthroplasty was performed for the first time （ 3) Good Chinese reading and comprehension ability （ 4) The patient's condition was stable, and there were no serious diseases of the heart, lung, brain and other important organs （ 5) Informed of the study and signed informed consent.

Exclusion Criteria:

（1）deep venous thrombosis of lower extremity （ 2) Other diseases affecting walking function （ 3) Suffering from cognitive or mental disorders （ 4) Had a history of knee surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients after total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-09-25 (Estimated); Study Completion 2021-09-25 (Estimated)

PRIMARY OUTCOMES:
The occurrence of fear of movement | 2nd day post-operative
  Score of Tampa for kinesiophobia(TSK) ranging from17-68.The higher score means the worse outcome

SECONDARY OUTCOMES:
Hospital Ansiety and Depression Scale(HADS) | 2nd day post-operative
  The score of HADS ranging from 0-48,the higher score means the worse outcome
General Self Efficacy Scale(GSES) | 2nd day post-operative
  The score of GSES,ranging from 1-40,the higher socre means the better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tao Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No